CLINICAL TRIAL: NCT04244422
Title: Clinical And Radiographic Outcomes Of Radicular Cyst Enucleation Using Piezosurgery Versus Conventional Surgery
Brief Title: Radicular Cyst Enucleation Using Piezosurgery Versus Conventional Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Gamaleldin Marei Noureldin, Lecturer of oral and maxillofacial surgery, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Piezosurgery cyst enucleation
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: RADICULAR CYSTS
MeSH Terms: conditions — Radicular Cyst

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyst enucleation using piezosurgery (Active Comparator): SATLEC ACTEON peizotome 2 was used for bone cutting and separating the cystic lining from the surrounding bone.After complete removal of the cyst, the bony window was replaced back in place and the flap was sutured.
  Interventions: Other: PIEZOSURGERY VERSUS CONVENTIONAL SURGERY
- cyst enucleation using conventional surgery (Active Comparator): A carbide bur was used to remove the bone to uncover the cyst. A periosteal elevator and a curette were used to aid in the removal of the cystic lesion.
  Interventions: Other: PIEZOSURGERY VERSUS CONVENTIONAL SURGERY

INTERVENTIONS:
Other: PIEZOSURGERY VERSUS CONVENTIONAL SURGERY — Piezosurgery: SATLEC ACTEON peizotome 2 (A company of ACTEON Group, France) was used. Conventional surgery with rotary instruments

SUMMARY:
AIM: The study was intended to evaluate the effectiveness of piezosurgery in enucleation of radicular odontogenic cysts in comparison to the conventional technique from both the clinical and radiographic perspectives.

DETAILED DESCRIPTION:
METHODS: Fourteen (8 females and 6 males) patients with age range of 30-55 years who had radicular cysts associated with non-vital teeth, were operated at the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University. The patients were randomly divided into 2 groups;1) the study group (7 patients) in which cyst enucleation using piezosurgery was employed, 2) control group in which the cysts were removed using the conventional technique. The following parameters were assessed; postoperative pain, time of operation, hemorrhage control and field visibility, ease of operation, neurosensory evaluation and radiographic percentage of change in bone defect volume between preoperative and 3-months postoperative values.

ELIGIBILITY:
Inclusion Criteria:

* 1) Periapical cysts involving more than one tooth in close relation to the maxillary sinus, nasal cavity or inferior alveolar neurovascular bundle,
* 2) Intact labial/buccal cortical plate with no perforation.

Exclusion Criteria:

* 1) Patients with systemic diseases contraindicating surgery
* 2) Cases in suspicion of malignancy

Ages: 31 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Time of operation in minutes | Intraoperative
  Time from start of the incision to the last suture.
Hemorrhage control and ease of operation using a visual analogue scale | Intraoperative
  To assess the visibility of the field and ease of operation, a visual analogue scale was used. Each parameter constituted a horizontal 100 mm continuous line in which value of zero indicates minimum level of the assessed parameter and 100 indicates the maximum level. Each surgeon marked on the line then the score is determined by measuring in mms from the left end of the line to that marked point. (higher scores mean a better outcome)
Objective assessment of neurosensory function using a probe (to detect nerve injury after the surgeries) | 1 month
  A probe was used to prick the patient's skin relevant to the area of operation to assess the neurosensory function in comparison to the contralateral side.If the patient states a difference in sensation between the side of operation and the normal side, it was assigned as "Y" and if there was no difference in sensation between the two sides, it was assigned as "N".
Radiographic percentage of change in bone defect volume using cone beam computed tomography | 3 months
  The change between preoperative and 3-months postoperative values of both groups were compared

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry-Alexandria University, Alexandria, Egypt